CLINICAL TRIAL: NCT01653275
Title: Mediterranean Diet for Post-menopausal Women: Effects on Bone Turnover
Acronym: MedSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Principal Investigator, Anne Kenny, Professor of Medicine, UConn Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-136S-1
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Osteoporosis; Postmenopausal Bone Loss
Keywords: Mediterranean Diet; Bone turnover; postmenopausal women
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mediterranean Diet (Experimental): Subjects will receive key foods (olive oil, walnuts, frozen portions of high n-3 LCPUFA fish) and instructed in the quantity to consume each week. Olive oil : minimum of 3 tablespoons per day. Walnuts:10.5 oz/week (1.5 oz/day). High n-3 LCPUFA fish: 3 or more fish meals per week. Additional guidelines for altering diet include incorporation of fruits, vegetables, legumes, and whole grains to replace sweets, white bread and starches, red meat and highly processed foods.
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Other: Mediterranean Diet — Subjects will receive key foods (olive oil, walnuts, frozen portions of high n-3 LCPUFA fish) and instructed in the quantity to consume each week. Olive oil : minimum of 3 tablespoons per day. Walnuts:10.5 oz/week (1.5 oz/day). High n-3 LCPUFA fish: 3 or more fish meals per week. Additional guidelines for altering diet include incorporation of fruits, vegetables, legumes, and whole grains to replace sweets, white bread and starches, red meat and highly processed foods.

SUMMARY:
The investigators propose a 24 week clinical research trial (12 week observational period followed by 12 week MedSD intervention) with feasibility of diet adoption and markers of bone turnover as the primary outcomes.

DETAILED DESCRIPTION:
Postmenopausal women are at increased risk of osteoporosis and fracture. Components of a Mediterranean style diet (MedSD) are associated with reduced bone loss and fracture risk; however, the MedSD has not been tested in this population in the U.S. Therefore, fhe investigators propose a 24 week clinical research trial (12 week observational period followed by 12 week MedSD intervention) with feasibility of diet adoption and markers of bone turnover as the primary outcomes. The 12 week intervention will include provision of olive oil, walnuts and high n-3 polyunsaturated fatty acids (PUFA) fish to replace other fats and oils, processed snacks and red meat, respectively; accompanied with fruit, vegetable, whole grain and legumes intake recommendations. The investigators hypothesize the MedSD intervention will increase serum n-3 PUFA and decrease saturated fatty acids and n-6 PUFA and this will result in an improvement in bone turnover markers. The outcomes of the proposed intervention trial will promote further study of the benefits of a MedSD in the US. the investigators envision the research team to expand to other systems such as cardiovascular, metabolic, and inflammatory mechanisms in which less risk of disease is associated with a MedSD.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women > 65 years
* BMI<30 kg/m2
* able to travel to clinical sites for follow-up visits
* willing to make no changes to habitual physical activity or calcium and vitamin D intake for the study duration

Exclusion Criteria:

* any disease that may affect bone metabolism, (i.e Paget's disease, primary hyperparathyroidism)
* cancers of any kind (except basal or squamous cell of skin) in past 5 years
* use of medication known to affect bone metabolism
* extreme dietary behaviors or supplementation in excess of DRI upper limits
* following a medically prescribed diet or dietary pattern similar to the MedSD
* history of chronic renal or liver disease
* history of hip fracture or known vertebral fracture within the past year
* persons with an allergy to fish or nuts.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
study adherence | 8 months
  Determine the extent to which postmenopausal women in the US can adhere to the MedSD intervention.

SECONDARY OUTCOMES:
Bone turnover markers | 8 months
  Determine if adherence to the MedSD will result in a reduction in bone resorption markers and enhance formation markers

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kenny, MD, Principal Investigator — UConn Health
Locations (1):
- UCHC, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided
only deidentified data will be available to share

REFERENCES:
- [Result] Bihuniak JD, Ramos A, Huedo-Medina T, Hutchins-Wiese H, Kerstetter JE, Kenny AM. Adherence to a Mediterranean-Style Diet and Its Influence on Cardiovascular Risk Factors in Postmenopausal Women. J Acad Nutr Diet. 2016 Nov;116(11):1767-1775. doi: 10.1016/j.jand.2016.06.377. Epub 2016 Aug 25. PMID 27568885